CLINICAL TRIAL: NCT03686891
Title: Analyis of the Prevalence of Sensitization to Legumes by Realistic Skin Prick Tests in a Patient Population Consulting at the University Hospital of Montpellier
Brief Title: Prevalence of Sensitization to Legumes in a Region From Southern France (Légumineuses)
Acronym: Légumineuses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 9776
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Sensitization to Legumes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Skin prick tests with four native legumes
  Interventions: Other: Skin prick tests with four native legumes

INTERVENTIONS:
Other: Skin prick tests with four native legumes — Skin prick tests with four native legumes

SUMMARY:
The Mediterranean diet is a model for health. Indeed, according to some epidemiological studies, it would participate in the prevention of various diseases such as cardiovascular diseases, diabetes type 2, cancer and obesity. Among the foods composing the Mediterranean diet, wheat and legumes are strongly represented. The introduction of legumes into an easily prepared and economical food for a large part of the population will lead to an increase in consumption. The combination of durum wheat semolina and legume flour would benefit from the nutritional qualities of the two raw materials (high protein, slow digestible carbohydrates, fiber, vitamins and minerals), but also of their double wheat-legume allergenicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in allergy consultation
* The patient (or parents for the under 18 years) must have given their free consent and signed the consent chart
* Men and women are included
* The patient is at least 2 years old

Exclusion Criteria:

* The patient is pregnant
* The patient is breast-feeding
* The patient is unable to stop in antihistamine medication for at least 7 days
* The patient refused or is unable to sign the consent chart
* The patient has a dermographism

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Sensitization rate to four cooked legumes in the population consulting in Allergy Unit at the University Hospital of Montpellier | 10 minutes (the average duration of the test will not be significantly increased)
  A prick test will be considered as positive in the presence of a wheal of urticaria of at least 3 mm in size

SECONDARY OUTCOMES:
Describe the population with positive skin prick tests to legumes | 5 years
  A prick test will be considered as positive in the presence of a wheal of urticaria of at least 3 mm in size
Associations between symptoms on ingestion of these legumes | 5 years
  Association between the positivity of the legume prick test and (1) symptoms upon ingestion of legumes (e.g., aracid and other fruits and vegetables), (2) symptoms of rhinitis, asthma, atopic eczema, and (3) positivity to other prick tests of the standard pneumallergen battery

CONTACTS AND LOCATIONS:
Locations (1):
- Service Exploration des allergologies-Hopital Arnaud de Villeneuve-CHU de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No